CLINICAL TRIAL: NCT01645189
Title: To Evaluate the Safety and Efficacy of Hunterase(Idursulfase-beta) in Hunter Syndrome Patients < 6 Years of Age Receiving Idursulfase Enzyme Replacement Therapy
Brief Title: Safety and Efficacy of Hunterase
Acronym: GC1111
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC1111C
Record Dates: First submitted 2012-07-16; First posted 2012-07-20 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hunter Syndrome
Keywords: Hunter syndrome; idursulfase-beta; Hunterase; GC1111
MeSH Terms: conditions — Mucopolysaccharidosis II

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test drug (Experimental): Idursulfase-beta
  Interventions: Biological: Hunterase

INTERVENTIONS:
Biological: Hunterase — once weekly, 0.5mg/kg IV infusion

SUMMARY:
The objective of this study is to determine the safety and efficacy of once weekly dosing of idursulfase-beta 0.5mg/kg administered by intravenous(IV) infusion for Hunter syndrome patients < 6 years old.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has a diagnosis of Hunter syndrome based upon biochemical criteria:

   * as measured in plasma, leukocytes, or fibroblasts,

     * a deficiency in iduronate-2-sulfatase (I2S) enzyme activity of ≤ 10 % of the lower limit of the normal range
   * That corresponds to one or more of the following:

     * a normal enzyme activity level of one other sulfatase
     * Confirmed as MPS2 by genetic test results
     * shows clinical symptoms/ visible signs of MPS2
2. < 6 years old and male
3. Patients who are able to comply with the study requirements
4. The patient's parent(s), or patient's legal guardian must have given voluntary written consent to participate in the study

Exclusion Criteria:

1. The patient has had a tracheostomy
2. The patient has known severe hypersensitivity or shock to any of the components of idursulfase
3. The patient has received treatment with another investigational therapy within 30 days prior to enrollment
4. History of a stem cell transplant
5. The patient has known severe hypersensitivity or shock to any of the components of test drug(excipient etc)

Max Age: 5 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | One year

SECONDARY OUTCOMES:
change of anti-idursulfase-beta antibody status | baseline and one year
Percent Change of Urine GAG | baseline to 53 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Kyu Jin, Principal Investigator — Samsung medical center, Seoul, Republic of Korea
Locations (1):
- Samsug Medical Center, Seoul, South Korea